CLINICAL TRIAL: NCT03062982
Title: A Phase I, Open-label, 2-sequence, Cross-over, Pharmacokinetic (PK) Study to Evaluate the Effect of the Food and to Identify the Metabolism of Fluzoparib in Healthy Subjects
Brief Title: Food-Effect and Metabolism Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FZPL-I-102-Food
Record Dates: First submitted 2017-02-09; First posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Solid Tumor
MeSH Terms: interventions — fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Administration of 120mg in fed state in Dosing Period 1 followed by administration of 120mg in fasted state in Dosing Period 2
  Interventions: Drug: Fluzoparib
- Group B (Experimental): Administration of 120mg in fasted state in Dosing Period 1 followed by administration of 120mg in fed state in Dosing Period 2
  Interventions: Drug: Fluzoparib

INTERVENTIONS:
Drug: Fluzoparib — 2 doses separated by 7 days.

SUMMARY:
This study evaluates the food-effect of one-dose Fluzoparib in healthy subjects. The participants receive Fluzoparib 120mg in fed state in Period 1 followed by administration of Fluzoparib 120mg in fasted state in Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent.
* Must be willing to comply with the requirements of the study.
* Willing to use a medically acceptable method (as defined by the Investigator) of birth control in the 6 months.
* Male or female aged 18-50 years.
* Weight more than 45kg, BMI within 18 and 28 kg/m2.
* No clinically significant abnormalities in physical examination and lab tests.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* No history of alcohol or drug abuse within the past year.
* Participation in any clinical trial of an experimental drug or device in the previous 3 months.
* Any medical condition or clinical laboratory test which in the judgment of the Investigator makes the subject unsuitable for the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | pre-dose and then 0.25、0.5、1、1.5、2、3、4、6、8、10、12、24、36、48、72、96h
  This study was designed to estimate the relative bioavailability of Fluzoparib 120 mg in the fed state relative to the fasted state.Peak Plasma Concentration (Cmax) and the the 90% confidence interval were calculated.
Pharmacokinetics-AUC | pre-dose and then 0.25、0.5、1、1.5、2、3、4、6、8、10、12、24、36、48、72、96h
  This study was designed to estimate the relative bioavailability of Fluzoparib 120 mg in the fed state relative to the fasted state.Area under the plasma concentration versus time curve (AUC0-last，AUC0-infinity) and the 90% confidence intervals were calculated.
Pharmacokinetics - Tmax (Hours) | pre-dose and then 0.25、0.5、1、1.5、2、3、4、6、8、10、12、24、36、48、72、96h
  To estimate the the time to Maximum concentration and constructe the corresponding 90% confidence intervals.
Collection of Feces and Urine and Measurement of 120mg Fluzoparib Metabolism in Healthy subjects by HPLC | 0-96h post dose if availabel
  This study was also designed to clarify the metabolism of Fluzoparib 120mg.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hosital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No